CLINICAL TRIAL: NCT05479786
Title: Evaluation of Reproductive Outcomes After Expectant or Surgical Management of a Previous Episode of Tubal Ectopic Pregnancy
Brief Title: Reproductive Outcomes After a Previous Episode of Tubal Ectopic Pregnancy in Patients Managed Expectantly and Surgically
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Collaborators: University of Debrecen (Other); Damascus University (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Palermo
Other Study IDs: ECTO-1
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic pregnancy; Expectant management; Pregnancy outcome; Salpingectomy; Salpingostomy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Watchful Waiting; Salpingectomy; Salpingostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ectopic pregnancy: Women with diagnosed tubal ectopic pregnancy
  Interventions: Other: Expectant management; Procedure: Salpingectomy; Procedure: Salpingostomy

INTERVENTIONS:
Other: Expectant management — Follow-up with beta-HCG dosages and transvaginal ultrasound scans
Procedure: Salpingectomy — Removal of the affected Fallopian tube by laparoscopy
Procedure: Salpingostomy — Removal of the ectopic pregnancy from the Fallopian tube, without removing the whole Fallopian tube, by laparoscopy

SUMMARY:
Although ectopic pregnancy was considered a leading cause of first-trimester maternal mortalities, current technological improvements allowed early diagnosis and opened a door for applying less invasive approaches. A tubal pregnancy could be managed either expectantly, medically, or surgically. The expectant management of ectopic pregnancy relies on the fact that a considerable proportion of ectopic gestations terminate by spontaneous tubal abortion. This approach is usually kept for stable cases with a small gestational sac and low beta-human chorionic gonadotropin (beta-HCG) serum levels. For hemodynamically unstable patients, higher levels of beta-HCG, and larger gestational sacs, surgery is often considered as the treatment of choice (16).

Considering this background, the study aims to analyze the subsequent natural reproductive outcomes of patients that had a previous tubal ectopic pregnancy and were managed either expectantly or surgically. Moreover, it amis to determine the factors that could influence the fertility potential of these patients in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Women with one episode of tubal ectopic pregnancy, treated by expectant management, salpingectomy, or salpingostomy;
* For patients treated surgically, only patients with at least one patent Fallopian tube confirmed via postoperative hysterosalpingography were included in the analysis.

Exclusion Criteria:

* Pregnancies of unknown location
* Other types of ectopic pregnancy
* Pelvic inflammatory disease
* Pelvic adhesions
* Intrauterine pathologies
* Pregnancies obtained after assisted-reproductive technologies (ART)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with either surgically-confirmed tubal ectopic pregnancy or a diagnosis of tubal ectopic pregnancy based on a positive beta-HCG serum measurement with the visualization of an adnexal mass resembling a tubal gestational sac and an empty uterine cavity upon transvaginal ultrasonographic scan.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Within one year after the previous episode of tubal ectopic pregnancy
  Presence of a gestational sac under ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — University of Palermo; Antoine Naem, M.D., Study Chair — Damascus University; Péter Török, M.D., Study Director — University of Debrecen

IPD SHARING:
Plan to Share IPD: Yes